CLINICAL TRIAL: NCT01450150
Title: Transcranial Direct Current Stimulation (tDCS) as an Augmenting Intervention for Treatment-Resistant Major Depression: A Randomized, Double-Blind and Sham-Controlled Trial
Brief Title: Transcranial Direct Current Stimulation as an Augmenting Intervention for Major Depression
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, MARCELO T. BERLIM, Director, Neuromodulation Research Clinic, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS-ERB08/04-2011
Record Dates: First submitted 2011-10-09; First posted 2011-10-12 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depression; Transcranial Direct Current Stimulation; Randomized, Sham-Controlled Trial; tDCS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — 20-minute daily sessions of 2 mA tDCS for 15 days (Monday to Friday on three consecutive weeks)
  Arms: Active tDCS
Device: Transcranial Direct Current Stimulation — The tDCS stimulator will be turned on for 30 seconds only, after which it will be gradually decreased and then turned off for the remainder of the 20-minute daily sessions for 15 days (Monday to Friday on three consecutive weeks).
  Arms: Sham tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is a noninvasive method to activate or de-activate neurons in superficial regions of the brain through the induction of weak electric currents in the brain tissue delivered by two scalp electrodes. Initial studies have shown tDCS to be effective for treating major depressive disorder (MDD), although there are negative trials in the specialized literature. One reason for these discrepant results might be that the duration of tDCS treatment in clinical trials to date (up to 2 weeks) is still insufficient to produce consistent clinical improvements. Thus, we intend to assess, in a sample of outpatients with MDD, whether a 3-week adjunctive course of active tDCS over the left dorsolateral prefrontal cortex is associated with a significant clinical improvement when compared to sham tDCS. The investigators hypothesize that subjects receiving active tDCS will present with significantly higher response and remission rates at weeks 3.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a current major depressive disorder (according to the Diagnostic and Statistical Manual, Fourth Edition, Text Revision [DSM-IV-TR])
* Baseline score ≥ 13 on the QIDS-C
* Stable medication regimen (> 4 weeks)

Exclusion Criteria:

* Psychotic features in the current episode
* Lifetime history of psychotic disorders and/or bipolar I or II disorders
* Substance or alcohol abuse/dependence in the past 6 months
* Lifetime history of a major neurological disease (e.g., Parkinson's, stroke)
* Uncontrolled medical disease (e.g., cardiovascular, renal)
* Pregnancy and/or lactation
* Presence of a specific contraindication for tDCS (e.g., personal history of epilepsy, metallic head implant, cardiac pacemaker)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory for Depressive Symptomatology - Clinician (QIDS-C) | week 4
  Response to treatment is defined as a ≥ 50% reduction in pretreatment symptoms severity at as measured by the mean QIDS-C score. Remission is defined as a QIDS-C score ≤ 5

SECONDARY OUTCOMES:
21-item Hamilton Depression Rating Scale (HAM-D21) | week 4
  Response to treatment is defined as a ≥ 50% reduction in the scores of the HAM-D21. Remission is defined as a HAM-D21 score ≤ 8
Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) | week 4
  Response is defined as a ≥ 50% reduction in the scores of the QIDS-SR. Remission is defined as a QIDS-SR score ≤ 5

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo T. Berlim, MD, MSc, Principal Investigator — McGill University & Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Nitsche MA, Boggio PS, Fregni F, Pascual-Leone A. Treatment of depression with transcranial direct current stimulation (tDCS): a review. Exp Neurol. 2009 Sep;219(1):14-9. doi: 10.1016/j.expneurol.2009.03.038. Epub 2009 Apr 5. PMID 19348793
- [Background] Murphy DN, Boggio P, Fregni F. Transcranial direct current stimulation as a therapeutic tool for the treatment of major depression: insights from past and recent clinical studies. Curr Opin Psychiatry. 2009 May;22(3):306-11. doi: 10.1097/YCO.0b013e32832a133f. PMID 19339889
- [Background] Arul-Anandam AP, Loo C. Transcranial direct current stimulation: a new tool for the treatment of depression? J Affect Disord. 2009 Oct;117(3):137-45. doi: 10.1016/j.jad.2009.01.016. Epub 2009 Feb 7. PMID 19201483
- [Background] Boggio PS, Rigonatti SP, Ribeiro RB, Myczkowski ML, Nitsche MA, Pascual-Leone A, Fregni F. A randomized, double-blind clinical trial on the efficacy of cortical direct current stimulation for the treatment of major depression. Int J Neuropsychopharmacol. 2008 Mar;11(2):249-54. doi: 10.1017/S1461145707007833. Epub 2007 Jun 11. PMID 17559710